CLINICAL TRIAL: NCT06230432
Title: Exploring the Mechanism of Severe Acute Pancreatitis Based on Metagenomics, Metabolomics and Proteomics
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Lingyu Luo, Professor, The First Affiliated Hospital of Nanchang University
Other Study IDs: FAH of NCU gastroenterology
Record Dates: First submitted 2023-12-29; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- healthy control
- mild acute pancreatitis
- moderately severe acute pancreatitis
- severe acute pancreatitis

SUMMARY:
The goal of this observational study is to learn about the biomarkers and mechanisms of severe acute pancreatitis in 30 healthy controls, 30 patients of mild acute pancreatitis, 30 patients of moderately severe acute pancreatitis, and 86 patients of severe acute pancreatitis. The main question it aims to answer are: • The relationship between changes in gut microbiota and clinical prognosis (plasma inflammatory cytokines, incidence and duration of infection in various parts, mortality rate), and the screening and validation of biomarkers that can be used for early prediction of disease severity. • Analyze the relationship between changes in blood composition and clinical prognosis (plasma inflammatory cytokines, incidence and duration of infection in various parts, mortality rate), screen and verify biomarkers that can be used for early prediction of disease severity. Blood and fecal samples from the healthy control group and diagnosed patients will be collected.

ELIGIBILITY:
Inclusion Criteria:

Patients group:

① Age between 18 and 75 years old;

② Within 72 hours of AP onset;

③ AP patients who meet the 2012 Atlanta AP Classification and Diagnostic Criteria.

Healthy control group:

* Age between 18 and 75 years old; ② No history of acute pancreatitis; ③ Routine laboratory tests such as blood routine and fecal routine are normal.

Exclusion Criteria:

* Used antibiotics, probiotics, and acid suppressants 4 weeks before enrollment;

  * Pregnant and lactating women;

    * Hypothyroidism, nephrotic syndrome, Cushing's syndrome, AIDS;

      * Chronic pancreatitis, pancreatic cancer; ⑤ Severe history of cardiovascular and cerebrovascular diseases and organ dysfunction, such as malignant tumors, heart failure, coronary heart disease, chronic obstructive pulmonary disease, liver and kidney failure; ⑥ Unsigned informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 healthy controls, 30 patients of mild acute pancreatitis, 30 patients of moderately severe acute pancreatitis and 86 patients of severe acute pancreatitis, a total of 176 cases were included.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2024-01-21 (Estimated); Primary Completion 2025-03-09 (Estimated); Study Completion 2026-12-09 (Estimated)

PRIMARY OUTCOMES:
Composition of gut microbiota | through study completion, an average of 1 year
  The gut microbiota plays an important role in protecting the intestinal barrier, regulating metabolism, and participating in immune responses in the human body, and is an important component of the gut ecosystem.
Composition of gut metabolites | through study completion, an average of 1 year
  Metabolites can reveal the intrinsic correlation between metabolic products and physiological and pathological changes in the body, thereby achieving recognition of the overall state of the body.
Composition of metabolites in plasma | through study completion, an average of 1 year
  Metabolites can reveal the intrinsic correlation between metabolic products and physiological and pathological changes in the body, thereby achieving recognition of the overall state of the body.
composition of proteins in plasma | through study completion, an average of 1 year
  Proteins are an important material foundation for life activities and the main executors of life processes such as cell proliferation, differentiation, aging, and death.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided